CLINICAL TRIAL: NCT05896787
Title: A Phase II Study of Candonilimab (AK104) Combined With Preoperative Chemotherapy in Patients With Locally Advanced Esophageal Squamous Cell Carcinoma (ESCC)
Brief Title: Candonilimab (AK104) Plus Preoperative Chemotherapy for Locally Advanced Esophageal Squamous Cell Carcinoma (ESCC)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Medical Oncology, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L2023-K003-002
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: AK104; preoperative chemotherapy; surgery
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — 130-nm albumin-bound paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104 plus nab-paclitaxel and carboplatin (Experimental): In the induction period, AK104 (10mg/kg, iv, Q2W) is given for one cycle;
  and then AK104 (10mg/kg, iv, Q3W) is combined with nab-paclitaxel (130mg/m2 ivgtt d1，d8, Q3W) and carboplatin ((AUC=5) d1，Q3W) for 2 cycles;
  After R0 surgery, AK104 (10mg/kg, iv, Q3W) is given as adjuvant therapy for up to 12 months for those who do not achieve pCR.
  Interventions: Drug: AK104, nab-paclitaxel, carboplatin

INTERVENTIONS:
Drug: AK104, nab-paclitaxel, carboplatin — AK104 plus nab-paclitaxel and carboplatin as neoadjuvant therapy，and AK104 as adjuvant therapy for those who do not achieve pCR;
  Other Names: Candonilimab，Preoperative Chemotherapy

SUMMARY:
This is a prospective, single-arm, open-label，multi-center, phase II study, aiming to evaluate the efficacy and safety of AK104 combined with preoperative chemotherapy in patients with locally advanced ESCC.

DETAILED DESCRIPTION:
Eligible patients first receive AK104 (10mg/kg, iv, Q2W) for one cycle in the induction period, and then patients receive AK104 (10mg/kg, iv, Q3W) combined with nab-paclitaxel (130mg/m2 ivgtt d1，d8, Q3W) and carboplatin ((AUC=5) d1，Q3W) for 2 cycles. After neoadjuvant therapy of 3 cycles, patient will undergo preoperative evaluation. For patients who can be performed for R0 surgery, surgery wil be performed in 4 to 6 weeks. Patients who do not achieve Pathological complete response (pCR) will receive AK104 (10mg/kg, iv, Q3W) as adjuvant therapy until disease progression or intolerable toxicity for up to 12 months. Patients who achieve pCR after surgery will be enrolled in observational follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signing a written informed consent form;
2. Males or females aged ≥ 18 to ≤ 70 years;
3. ECOG score 0-1;
4. Pathologically diagnosed thoracic esophageal squamous cell carcinoma;
5. No distant metastasis after imaging examination, and esophageal cancer can be resected or potentially resectable with stage cT1b-cT2N+M0 or cT3-cT4a anyN M0 or cT2N0M0 high-risk (lymphovascular invasion or tumor ≥3 cm or hypo-differentiation) (AJCC 8th edition cTNM stage);
6. Not received prior antitumor therapy (surgery, radiotherapy, chemotherapy, immunotherapy, etc. for esophageal cancer);
7. Life expectancy is greater than 6 months;
8. At least one measurable tumor lesion per RECIST v1.1;
9. Major organ functions are adequate;

Exclusion Criteria:

1. Patient has received previous antitumor therapy (chemotherapy, radiation, surgery or immunotherapy);
2. Cervical or thoracic esophageal cancer is < 5 cm from the cricopharyngeal muscle;
3. Patients are or are expected to be at significant risk of esophageal perforation, fistula, and major bleeding;
4. Imaging during the screening period showed that the tumor surrounded or invaded important blood vessels or organs (such as the heart and pericardium, trachea, aorta, superior vena cava, etc.) or there was obvious necrosis or cavity, and the investigator determined that entering the study would cause bleeding risk; participants at risk of developing oesophageal or oesophageal fistula;
5. Patients with a history of other malignant diseases in the last 5 years，unless complete resolution or no additional treatment is required (exceptions include, but are not limited to, basal or squamous cell skin cancer, superficial bladder cancer or prostate, cervix, or breast carcinoma in situ)；
6. Pregnant or nursing women；
7. Patients with known or suspected active autoimmune disease;
8. Patients with a history of myocarditis, cardiomyopathy, malignant arrhythmias;
9. Other patients are not eligible for enrollment assessed by investigators;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
pCR | up to 2 years
  Pathological complete response

SECONDARY OUTCOMES:
MPR | up to 2 years
  Major pathologic response
R0 resection rate | up to 2 years
  R0 resection rate
Downstaging rate | up to 2 years
  Downstaging rate
DFS | up to 2 years
  Disease-free survival
OS | up to 2 years
  Overall survival
AE | up to 2 years
  Adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (2):
- China (2):
  - Anyang Cancer Hospital, Anyang, Henan
  - Feng Wang, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No